CLINICAL TRIAL: NCT07302347
Title: A Phase I/II Study of Pembrolizumab (MK-3475) in Japanese Pediatric Participants With Specific Solid Tumors or Lymphomas, or in Japanese Adult Participants With Advanced Merkel Cell Carcinoma (KEYNOTE-G21)
Brief Title: A Study of Pembrolizumab in Japanese Pediatric Participants With Solid Tumors or Lymphomas and Japanese Adult Participants With Merkel Cell Carcinoma (MK-3475-G21/KEYNOTE-G21)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-G21; MK-3475-G21 (Other: MSD)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasm; Carcinoma, Merkel Cell; Lymphoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Merkel Cell; Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: No blinding for Arm 1. Outcomes assessor blinded for Arm 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pembrolizumab in Pediatric Participants with Solid Tumors or Lymphomas (Experimental): Pediatric participants with solid tumors or lymphomas receive 2 mg/kg pembrolizumab via intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21 day cycle for up to 17 or 35 cycles.
  Interventions: Biological: Pembrolizumab
- Arm 2: Pembrolizumab in Adult Participants with Merkel Cell Carcinoma (MCC) (Experimental): Adult participants with MCC receive 400 mg pembrolizumab via IV infusion on Day 1 of each 42 day (6 week) cycle, for up to 18 cycles.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — 25 mg/mL solution for intravenous infusion.
  Other Names: MK-3475

SUMMARY:
Researchers are looking for new ways to treat people with solid tumors, lymphomas (blood cancers), and a certain type of skin cancer. The goals of this study are to learn:

* About the safety of pembrolizumab (the study medicine) and if people tolerate it
* What happens to different doses of pembrolizumab in a person's body over time
* How the cancer responds (gets smaller or goes away) to treatment

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

Arm 1:

* For participants with relapsed or refractory classical Hodgkin lymphoma (cHL) or primary mediastinal large B-cell lymphoma (PMBCL)

  * Has a confirmed diagnosis of relapsed or refractory cHL or PMBCL after the most recent therapy
  * Has radiographically measurable disease per Lugano classification
* For participants with completely resected melanoma:

  * Has surgically completely resected and histologically/pathologically confirmed diagnosis of Stage IIB, IIC, III or IV cutaneous melanoma
  * Has not received any prior systemic therapy for their melanoma beyond surgical resection
  * All suspicious lesions amenable to biopsy are confirmed negative for malignancy
* For participants with locally advanced or metastatic melanoma:

  * Has histologically confirmed diagnosis of locally advanced (unresectable Stage III) or metastatic (Stage IV) melanoma (including acral) not amenable to local therapy
  * Has radiographically measurable lesion(s) as defined by RECIST 1.1
* For participants with microsatellite instability-high (MSI-H)/mismatch repair deficiency (dMMR) solid tumors:

  * Has histologically/cytologically documented, locally-advanced, or metastatic solid malignancy that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the participant and treating physician
  * Has a documented positive local MSI-H or dMMR test result
  * Has radiographically measurable disease based on RECIST 1.1
* For participants with tumor mutational burden-high (TMB-H) solid tumors:

  * Has histologically/cytologically documented, locally-advanced, or metastatic solid malignancy that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the participant and treating physician
  * Has radiographically measurable disease based on RECIST 1.1
* For participants with MCC:

  * Has histologically confirmed diagnosis of locoregional MCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy and is not amenable to local therapy or metastatic MCC (Stage IV)
  * Has radiographically measurable disease based on RECIST 1.1

Arm 2:

* For participants with MCC:

  * Has been untreated for advanced or metastatic disease

Arm 1 & Arm 2:

* Life expectancy of >3 months (Arm 1) or >6 months (Arm 2)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has known additional malignancy that is progressing or has required active treatment
* Has known active (central nervous system) CNS metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in past 2 years
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV) infection
* Has known history of Hepatitis B infection or known active Hepatitis C virus
* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic stem cell transplantation within the last 5 years
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Arm 1: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 28 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. The number of participants with solid tumors or lymphomas who experience an AE will be reported.
Arm 1: Number of Participants Who Discontinue Study Treatment Due To an AE | Up to approximately 25 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. The number of participants with solid tumors or lymphomas who discontinue study treatment due to an AE will be reported.
Arm 1: Area Under the Concentration-Time Curve (AUC) of Pembrolizumab | Predose at Cycle 1, 2, 4, 8 and every 4 cycles thereafter up to 35 cycles; postdose at Cycle 1 and Cycle 8 (a cycle is 21 days)
  AUC is defined as the area under the concentration-time curve of pembrolizumab. Blood samples will be collected at specified intervals for the determination of AUC. AUC in participants with solid tumors or lymphomas will be reported.
Arm 1: Maximum Concentration (Cmax) of Pembrolizumab | Predose at Cycle 1, 2, 4, 8 and every 4 cycles thereafter up to 35 cycles; postdose at Cycle 1 and Cycle 8 (a cycle is 21 days)
  Cmax is defined as the maximum concentration of pembrolizumab reached. Blood samples will be collected at pre-specified intervals for the determination of Cmax. Cmax in participants with solid tumors or lymphomas will be reported.
Arm 1: Minimum Plasma Concentration (Cmin) of Pembrolizumab | Predose at Cycle 1, 2, 4, 8 and every 4 cycles thereafter up to 35 cycles; postdose at Cycle 1 and Cycle 8 (a cycle is 21 days)
  Cmin is defined as the minimum concentration of pembrolizumab observed in plasma after its administration and just prior to administration of a subsequent dose. Blood samples will be collected at pre-specified timepoints to determine Cmin. Cmin in participants with solid tumors or lymphomas will be reported.
Arm 2: Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) | Up to approximately 37 months
  ORR is defined as complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by blinded independent central review (BICR). ORR in participants with Merkel cell carcinoma will be reported.

SECONDARY OUTCOMES:
Arm 1: ORR per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  ORR is defined as complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by investigator assessment. ORR in participants with solid tumors will be reported.
Arm 1: ORR per Lugano Classification by Investigator Assessment | Up to approximately 46 months
  ORR is defined as complete response (CR: all target lymph nodes must have regressed to normal size defined as ≤1.5 cm in longest diameter) or partial response (PR: ≥50% decrease in sum of products of diameters of target lesions from baseline, and no individual lesion meets the criteria for progression), per Lugano classification (Cheson et al, Journal of Clinical Oncology, 2014). ORR in participants with lymphomas as assessed by investigator will be reported.
Arm 1: Duration of Response (DOR) per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  For participants who demonstrate a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR per RECIST 1.1 by investigator assessment in participants with solid tumors will be reported.
Arm 1: DOR per Lugano Classification by Investigator Assessment | Up to approximately 46 months
  For participants who demonstrate confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR (all target lymph nodes must have regressed to normal size defined as ≤1.5 cm in longest diameter) or PR (≥50% decrease in sum of products of diameters of target lesions from baseline, and no individual lesion meets the criteria for progression) per Lugano classification (Cheson et al, Journal of Clinical Oncology, 2014) until progressive disease (PD: based on the progression of any single lesion and other certain requirements) or death due to any cause, whichever occurs first. DOR in participants with lymphomas as assessed by investigator will be reported.
Arm 1: Disease Control (DCR) per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR or PR or stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]). DCR per RECIST 1.1 by investigator assessment in participants with solid tumors will be reported.
Arm 1: DCR per Lugano Classification by Investigator Assessment | Up to approximately 46 months
  DCR is defined as confirmed CR (all target lymph nodes must have regressed to normal size defined as ≤1.5 cm in longest diameter), PR (≥50% decrease in sum of products of diameters of target lesions from baseline, and no individual lesion meets the criteria for progression), or stable disease (SD: Target lesions do not meet the criteria for CR or PR and no individual lesion meets the criteria for progression) per Lugano classification (Cheson et al, Journal of Clinical Oncology, 2014). DCR in participants with lymphomas as assessed by investigator will be reported.
Arm 1: Progression-free Survival (PFS) per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS per RECIST 1.1 by investigator assessment in participants with solid tumors will be reported.
Arm 1: PFS per Lugano Classification by Investigator Assesment | Up to approximately 46 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Lugano classification (Cheson et al, Journal of Clinical Oncology, 2014) by investigator. PD per Lugano classification is defined as based on the progression of any single lesion and other certain requirements. PFS in participants with solid tumors will be reported.
Arm 1: Relapse-free Survival (RFS) per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  RFS is defined only for adjuvant melanoma participants as the time from first dose to recurrence of melanoma at any site (local, in-transit or regional lymph nodes or distant recurrence) per RECIST 1.1 by investigator assessment or death due to any cause, whichever occurs first. New incident cases of melanoma and second cancer diagnoses are not counted as events for recurrence-free survival. RFS in participants with solid tumors or lymphomas will be reported.
Arm 1: Distant Metastasis-free Survival (DMFS) per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  DMFS is defined only for adjuvant melanoma participants as the time from first dosing to the first diagnosis of a distant metastasis per RECIST 1.1 by investigator assessment or death (due to any cause), whichever occurs first. Distant metastasis refers to cancer that has spread from the original (primary) tumor and beyond local tissues and lymph nodes to distant organs or distant lymph nodes. DMFS in participants with solid tumors or lymphomas will be reported.
Arm 1: Overall Survival (OS) | Up to approximately 46 months
  OS is defined as the time from the first dose of study intervention to death due to any cause. OS in participants with solid tumors or lymphomas will be reported.
Arm 1: Number of Participants with Anti-Drug Antibodies (ADAs) Against Pembrolizumab | Predose at Cycle 1, 2, 4, 8 and every 4 cycles thereafter up to 35 cycles (a cycle is 21 days)
  Blood samples will be collected at multiple time points to determine the ADA response to pembrolizumab. The number of participants with ADA for pembrolizumab in participants with solid tumors or lymphomas will be reported.
Arm 2: ORR per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  ORR is defined as complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by investigator assessment. ORR in participants with Merkel cell carcinoma will be reported.
Arm 2: DOR per RECIST 1.1 by BICR | Up to approximately 46 months
  For participants who demonstrate a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR per RECIST 1.1 by BICR in participants with Merkel cell carcinoma will be reported.
Arm 2: DOR per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  For participants who demonstrate a confirmed CR: disappearance of all target lesions or PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR by investigator assessment in participants with Merkel cell carcinoma will be reported.
Arm 2: DCR per RECIST 1.1 by BICR | Up to approximate ly 46 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR or PR or stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]). DCR per RECIST 1.1 by BICR in participants with Merkel cell carcinoma will be reported.
Arm 2: DCR per RECIST 1.1 by Investigator Assessment | Up to approximately 46 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR or PR or stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD). DCR per RECIST 1.1 by investigator assessment in participants with Merkel cell carcinoma will be reported.
Arm 2: PFS per RECIST 1.1 by BICR | Up to approximately 46 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS per RECIST 1.1 by BICR in participants with Merkel cell carcinoma will be reported.
Arm 2: PFS per RECIST 1.1 by Investigator Assesment | Up to approximately 46 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS per RECIST 1.1 by investigator assessment in participants with Merkel cell carcinoma will be reported.
Arm 2: OS | Up to approximately 46 months
  OS is defined as the time from the first dose of study intervention to death due to any cause. OS in participants with Merkel cell carcinoma will be reported.
Arm 2: Cmax of Pembrolizumab | Predose at Cycles 1-4, and every 2 cycles thereafter up to 18 cycles; postdose at Cycle 1 and Cycle 3 (a cycle is 42 days)
  Cmax is defined as the maximum concentration of pembrolizumab reached. Blood samples will be collected at pre-specified intervals for the determination of Cmax. Cmax in participants with Merkel cell carcinoma will be reported.
Arm 2: Cmin of Pembrolizumab | Predose at Cycles 1-4, and every 2 cycles thereafter up to 18 cycles; postdose at Cycle 1 and Cycle 3 (a cycle is 42 days)
  Cmin is defined as the minimum concentration of pembrolizumab observed in plasma after its administration and just prior to administration of a subsequent dose. Blood samples will be collected at pre-specified timepoints to determine Cmin. Cmin in participants with Merkel cell carcinoma will be reported.
Arm 2: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 28 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. The number of participants with Merkel cell carcinoma who experience an AE will be reported.
Arm 2: Number of Participants Who Discontinue Study Treatment Due To an AE | Up to approximately 25 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study intervention. The number of participants with Merkel cell carcinoma who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/